CLINICAL TRIAL: NCT02289079
Title: Ultrasound Guided Subcostal Transversus Abdominis Plane (TAP) Block With Liposomal Bupivacaine vs Bupivacaine in Robotic Hysterectomy Patients: A Prospective Randomized Study.
Brief Title: TAP Block With Liposomal Bupivacaine Versus Bupivacaine in Robotic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1305m34041
Record Dates: First submitted 2014-10-30; First posted 2014-11-13 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- liposomal bupivacaine TAP (Experimental): these patients receive a subcostal TAP with liposomal bupivacaine
  Interventions: Drug: liposomal bupivacaine
- bupivacaine TAP (Active Comparator): These patients receive a subcostal TAP with bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine
  Arms: bupivacaine TAP
Drug: liposomal bupivacaine
  Arms: liposomal bupivacaine TAP

SUMMARY:
The purpose of the study is to compare pain control after robotic hysterectomy surgery using either liposomal bupivacaine or Bupivacaine when injected during a transversus abdominis plane (TAP) block. Robotic hysterectomy is when a patient is electively having robotic assisted removal of one's uterus. Both medications liposomal bupivacaine and Bupivacaine are standard of care in these types of surgeries.

DETAILED DESCRIPTION:
Treatment technique:

The patient will be in the supine position. The transversus abdominis muscle layer will be identified with the ultrasound. Using sterile technique, skin infiltration with 2% lidocaine will occur, 2 cm medial to the ultrasound probe. An 22g Nerve block needle will then be inserted and advanced under ultrasound guidance until it is below the fascial covering of the transversus abdominis muscle layer. Gentle aspiration for air, or blood will be performed and either 30 cc of 0.25% bupivacaine with 1/200,000 parts epinephrine or 30 mL of liposomal bupivacaine mixed 1:1 with normal saline will be injected under ultrasound guidance. For each 5cc of local anesthetic injected, aspiration will be performed. Upon completion of the injection, the needle will then be removed. This will then be completed on the contralateral side. The patient will be monitored in the preoperative area until he/she is brought into the operating room for their procedure.

When the operation is complete the patient will either be discharged home or brought to the ward where each day a member of the research team will evaluate the patient for signs of complications and ask the patient their minimum and maximum pain score.

If patients have met criterion for discharge to home including pain <4/10, independence of intravenous analgesia, and are stable for discharge medically, but are awaiting placement, the time of discharge for the purposes of the study will be the day they have met such criterion as opposed to the day of actual discharge, as this can vary depending on patient placement.

If the patient is discharged prior to 72 hours post injection, then the patient will receive one phone call at 24 hours post injection, 48 hours post injection , and 72 hours post injection +/- 5 hours. During this phone call the patient will be asked about pain score, narcotic use, overall satisfaction via a recorded patient questionnaire, quality of recovery via a quality of recovery survey, and assessed if any adverse events have occurred.

Adequate analgesia will be defined as <3 VAS at rest, and if VAS is greater than 3 adjustments in oral or intravenous pain medications will be given as determined by the nurse.

ELIGIBILITY:
Inclusion Criteria:

* those who present for elective robotic assisted hysterectomy

Exclusion Criteria:

* non english speaking
* chronic pain
* on opioids greater than 1 weeks
* chronic anticoagulation
* allergy to local anesthetics
* use of spinal or epidural for surgery
* lack of patient cooperation
* contraindication to regional anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

REFERENCES:
- [Derived] Hutchins J, Delaney D, Vogel RI, Ghebre RG, Downs LS Jr, Carson L, Mullany S, Teoh D, Geller MA. Ultrasound guided subcostal transversus abdominis plane (TAP) infiltration with liposomal bupivacaine for patients undergoing robotic assisted hysterectomy: A prospective randomized controlled study. Gynecol Oncol. 2015 Sep;138(3):609-13. doi: 10.1016/j.ygyno.2015.06.008. Epub 2015 Jun 6. PMID 26056753

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine TAP: these patients receive a subcostal TAP with liposomal bupivacaine
  liposomal bupivacaine
- Bupivacaine TAP: These patients receive a subcostal TAP with bupivacaine
  Bupivacaine
Period: Overall Study
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Started | 30 | 30
Completed | 28 | 29
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 25 | 45
  >=65 years | 8 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 58
weight [Mean (Standard Deviation); unit: kilograms] | 89.3 (25.1) | 98.5 (34.2) | 93.5 (30.2)

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Opioid Use
Description: To determine if liposomal bupivacaine provides decreased narcotic use when compared to bupivacaine when injected in a TAP block
Time Frame: 0-72 hours after injection
Measure: Median (Full Range); unit: micrograms of fentanyl equivalents
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Number analyzed (Participants) | 28 | 29
micrograms of fentanyl equivalents | 24.9 [0 to 86.7] | 51.7 [0 to 249.7]

2. Secondary Outcome: Numerical Rating Scale
Description: This was a measure of patient's reported pain on a 0-10 verbal numerical rating scale. 10 being worst pain. The maximal value for the time period 48-72 hours was chosen as the maximal pain during that time period.
Time Frame: 48-72 hours
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Number analyzed (Participants) | 28 | 29
scores on a scale | 3 [0 to 8] | 5 [0 to 10]

3. Secondary Outcome: Post Operative Length of Stay
Description: To determine if liposomal bupivacaine provides decreased length of stay when compared to bupivacaine when injected in a TAP block
Time Frame: up to 30 days after surgery
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Number analyzed (Participants) | 28 | 29
Hours | 11 (9.1) | 17 (13.9)

4. Secondary Outcome: Patient Satisfaction as Assessed Via Patient Survey
Description: To determine if liposomal bupivacaine improves quality of recovery post-operatively when compared to bupivacaine when injected in a TAP block via a patient survey either in person or via telephone.
Time Frame: assessed at 72 hours after injection
Measure: Number; unit: participants satisfied with pain control
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Number analyzed (Participants) | 28 | 29
participants satisfied with pain control | 26 | 24

ADVERSE EVENTS:
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes